CLINICAL TRIAL: NCT02717078
Title: A Weight Neutral, High Protein, Moderate Carbohydrate Diet for Treatment of Type 2 Diabetes Mellitus
Brief Title: The LoBAG Diet and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2016-23735
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diet; carbohydrate; protein; glucose; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LoBAG Diet (Experimental): Assignment to consume the LoBAG diet (30% carbohydrate, 30% protein, 40% fat; carbohydrates that are low in starch emphasized) for 12 weeks.
  Interventions: Other: Diet Therapy
- Control Diet (Active Comparator): Assignment to consume the control diet (50% carbohydrate, 15% protein, 35% fat) for 12 weeks.
  Interventions: Other: Diet Therapy

INTERVENTIONS:
Other: Diet Therapy — The intervention for both study groups will be a change in diet.

SUMMARY:
The proposed study is a randomized controlled, pilot effectiveness trial comparing the LoBAG diet to a control diet in 38 participants with DM2 over 12 weeks. Participants will have DM2 that is not under ideal glycemic control (HgbA1c 7.0-9.5%) and must be taking no glycemic medications or metformin. Participants will be free-living (given diet instruction and dietitian support, but asked to prepare meals in their own homes). The primary endpoint will be HgbA1c, measured at baseline and at the end of the 12-week diet intervention. Additional outcome measures will include: weight, fasting plasma glucose, fasting serum insulin, postprandial plasma glucose and serum insulin following a test meal consistent with the assigned diet, serum fructosamine, fasting serum lipids, stool samples for gut microbiome analysis, and surveys to assess quality of life, including the Diabetes Treatment Satisfaction Questionnaire. Compliance outcomes will include: urine nitrogen to creatinine ratio, survey data, three-day food diaries, and unannounced 24-hour diet recalls.

DETAILED DESCRIPTION:
Thirty-eight adult men and women with DM2 will be recruited from the University of Minnesota and surrounding communities, and will be randomized to treatment with the LoBAG diet or a control diet. Following a consent and screening visit, there will be 5 additional study visits over a 12-week diet intervention period. Instruction in the assigned diet will be provided by a research dietitian at the beginning of the 12-week period, and reinforced at subsequent visits throughout the study. Participants will be asked to purchase food, prepare food, and consume the assigned diet in their own homes. They will be asked to keep activity level constant and to continue medications for diabetes (metformin or no medication) without change during the intervention. The primary outcome, HgbA1c, and secondary outcome measures will be assessed at baseline and following diet intervention. Study visits will occur at baseline (visits 1 and 2), week 1 (visit 3), week 6 (visit 4), week 9 (visit 5) and week 12 (final study visit). In addition to scheduled study visits the research team will contact participants every other week by telephone to address any issues that arise, with the purpose of increasing compliance and retention. Participants will be contacted once in weeks 9-12 for a 24-hour diet recall collected by the Nutrition Coordinating Center at the University of Minnesota. Study procedures will conclude after the 12-week diet intervention period and collection of all outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of type 2 diabetes mellitus
* Hemoglobin A1c of 7.0-9.5%
* Taking no medications for diabetes or taking metformin

Exclusion Criteria:

* Type 1 diabetes mellitus
* Treatment with insulin
* BMI < 27 kg/m^2
* Change in weight of more than 5 pounds in the prior 3 months
* Estimated glomerular filtration rate (GFR) < 60 ml/minute/1.73 m^2
* Urine albumin > 300 mg/g creatinine
* Anemia
* Pregnancy or immediate plans to become pregnant
* Current breast feeding
* Use of antibiotics in the 3 month period prior to study enrollment
* Dietary restriction(s) that would preclude consumption of the study diets
* Inability or unwillingness to prepare meals
* Presence of any disease which would make adherence to the study protocol difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Bantle, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LoBAG Diet | Control Diet
Started | 24 | 24
Completed | 20 | 18
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LoBAG Diet | Control Diet | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.1) | 55.8 (11.5) | 57.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 30
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 21 | 16 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c From Baseline to Week 12
Description: Marker of blood sugar control
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | LoBAG Diet | Control Diet
Number analyzed (Participants) | 20 | 18
percentage | 6.6 (0.6) | 7.2 (0.8)

2. Secondary Outcome: Change in Weight From Baseline to Week 12
Description: Weight in pounds
Time Frame: Week 12
Reporting Status: Not Posted

3. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 12
Description: Blood draw
Time Frame: Week 12
Reporting Status: Not Posted

4. Secondary Outcome: Change in Fasting Serum Insulin From Baseline to Week 12
Description: Blood draw
Time Frame: Week 12
Reporting Status: Not Posted

5. Secondary Outcome: Postprandial Plasma Glucose and Serum Insulin Following a Test Meal
Description: A meal will be provided, and blood drawn at regular intervals for 4 hours following the meal
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Postprandial Plasma Glucose and Serum Insulin Following a Test Meal
Description: A meal will be provided, and blood drawn at regular intervals for 4 hours following the meal
Time Frame: Week 12
Reporting Status: Not Posted

7. Secondary Outcome: Change in Serum Fructosamine From Baseline to Week 12
Description: A marker of blood sugar control, similar to hemoglobin A1c
Time Frame: Week 12
Reporting Status: Not Posted

8. Secondary Outcome: Change in Fasting Serum Lipids From Baseline to Week 12
Description: Blood draw
Time Frame: Week 12
Reporting Status: Not Posted

9. Secondary Outcome: Diabetes Treatment Satisfaction Questionnaire Score
Description: Questionnaire to determine satisfaction with current diabetes treatment, scored 0 (very dissatisfied) to 36 (very satisfied)
Time Frame: Week 12
Reporting Status: Not Posted

10. Secondary Outcome: Gut Microbiome Composition
Description: The human gut microbiome refers to the bacteria, fungi, and viruses that inhabit the human intestine. Participants will be asked to collect a small sample of stool on a swab. Collection will be done at home.
Time Frame: Baseline
Reporting Status: Not Posted

11. Secondary Outcome: Gut Microbiome Composition
Description: as for outcome 10
Time Frame: Week 6
Reporting Status: Not Posted

12. Secondary Outcome: Gut Microbiome Composition
Description: as for outcome 10
Time Frame: Week 12
Reporting Status: Not Posted

13. Secondary Outcome: Urine Nitrogen to Creatinine Ratio
Description: Urine sample
Time Frame: Baseline
Reporting Status: Not Posted

14. Secondary Outcome: Urine Nitrogen to Creatinine Ratio
Description: Urine sample
Time Frame: Week 3
Reporting Status: Not Posted

15. Secondary Outcome: Urine Nitrogen to Creatinine Ratio
Description: Urine sample
Time Frame: Week 6
Reporting Status: Not Posted

16. Secondary Outcome: Urine Nitrogen to Creatinine Ratio
Description: Urine sample
Time Frame: Week 9
Reporting Status: Not Posted

17. Secondary Outcome: Urine Nitrogen to Creatinine Ratio
Description: Urine sample
Time Frame: Week 12
Reporting Status: Not Posted

18. Secondary Outcome: Three-day Food Diary
Description: Meal record for 3 days
Time Frame: Baseline
Reporting Status: Not Posted

19. Secondary Outcome: Three-day Food Diary
Description: Meal record for 3 days
Time Frame: Week 6
Reporting Status: Not Posted

20. Secondary Outcome: Three-day Food Diary
Description: Meal record for 3 days
Time Frame: Week 12
Reporting Status: Not Posted

21. Secondary Outcome: 24-hour Diet Recall
Description: Interview to review meals consumed in previous 24 hours
Time Frame: Week 9
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | LoBAG Diet | Control Diet
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 3/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LoBAG Diet (N=24) | Control Diet (N=24)
Nausea (General disorders) | 1 (1) | 0 (0)
tingling/neuropathy symptoms (Nervous system disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
arm pain (General disorders) | 0 (0) | 1 (1) — not related to CGM sensor
kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1)
back injury (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT02717078/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/78/NCT02717078/ICF_001.pdf